CLINICAL TRIAL: NCT05281393
Title: PrEP2Prevent: An Online PrEP Navigation and Activation Intervention for YMSM, Trans and Non-Binary Youth (PrEP2Prevent HIV)
Brief Title: PrEP2Prevent An Online PrEP Navigation and Activation Intervention
Acronym: P2P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Florida State University (Other)
Responsible Party: Principal Investigator, Michele D. Kipke, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHLA-20-00596
Record Dates: First submitted 2022-01-06; First posted 2022-03-16 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: HIV Infections
Keywords: PrEP; Mobile Health; LGBTQ; Transgender; Adolescent
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Access to mobile health platform for resources and information about PrEP
- Experimental (Experimental): Access to mobile health platform for resources and information about PrEP plus sessions with peer health support navigator, social app interactions, goal setting capabilities
  Interventions: Behavioral: PrEPresent

INTERVENTIONS:
Behavioral: PrEPresent — PrEP2Prevent is being done in several phases (parts) to develop and pilot test a PrEP activation, navigation and support intervention for young men who have sex with men (YMSM), trans youth and non-binary youth in Los Angeles. It targets an intervention for these young people where they need it most - on PrEP uptake. PrEP stands for pre-exposure prophylaxis.
  Other Names: PrEP2Prevent
  Arms: Experimental

SUMMARY:
* The goal of this clinical trial entitled, PrEP2Prevent: An Online PrEP Navigation and Activation Intervention for YMSM, is to develop and test a method for supporting access to an HIV prevention medication called Pre-Exposure Prophylaxis (PrEP) in young men who have sex with men and young transgender and non-binary individuals. The main questions it aims to answer are:
* What are some of the experiences and barriers providers have seen regarding this population accessing PrEP
* Using information gathered from PrEP providers and navigators, develop a mobile health platform and PrEP related content that will be tested by members of the population to see if the features are usable and the content is understandable.
* Enroll 150 study participants to see if utilizing the mobile health platform and receiving supportive sessions related to motivation and barriers to accessing PrEP is achievable.
* Participants will
* Be given access to the mobile health Platform called PrEPresent, which provides them with access to prevention related content, the ability to schedule with a patient navigator and create customizable goals
* Complete a baseline, 3 month and 6 month assessment about personal health, health history and technology, along with a PrEP adherence rapid urine test
* Complete up to 4 sessions to assist participants in the intervention group with discussing any barriers to accessing PrEP

DETAILED DESCRIPTION:
The U.S. Department of Health and Human Services (HHS) has set a goal to end the HIV epidemic by the year 2030, which is well within reach given the availability of antiretrovirals that effectively prevent and treat HIV. But success can only be achieved if targeted approaches are implemented with at-risk populations to address known barriers of engagement along the pre-exposure prophylaxis (PrEP) and HIV care continua. In response, obtained funding from NIH, using the R34 mechanism, with the goal of the research being to develop and pilot test a PrEP activation, navigation and support intervention for YMSM, including young Black and Latino YMSM (B-YMSM, L-YMSM), who not only have the highest annual incidence of HIV but who are also the least likely to have ever used PrEP. There is very clear evidence demonstrating that while YMSM have high levels of knowledge about and intentions to use PrEP, few have ever used PrEP. Our own research demonstrate the urgent need for interventions that specifically target PrEP uptake while also addressing a complex array of individual (e.g., side effect concerns, substance use, depression), sociocultural (e.g., internalized homophobia, PrEP-related stigma), and structural (e.g., access to care, medication costs) barriers to PrEP uptake. Our research also demonstrates that such an intervention should include four components: 1) inclusion of PrEP and other service navigation; 2) provision of skills to address patient activation, reduce PrEP-related stigma, and increase PrEP self-efficacy; 3) peer/social support; and 4) utilize a mobile health (mHealth) platform or similar technology that supports both in-person and virtual intervention delivery (text and live video chat). Based on these findings, the investigators propose to conduct research with the following specific aims

Specific Aim 1: Conduct formative research to inform the development of a PrEP activation, navigation and support intervention, which the investigators call PrEP2Prevent. Qualitative data will be collected using structured guides from working/focus groups with YMSM, Trans, and gender non-conforming youth and during Key Informant Interviews (KII) with existing PrEP care providers/navigators. These data will inform intervention content and activation/navigation services.

Specific Aim 2: Develop and then conduct usability testing of PrEP2Prevent, including both the intervention content and mHealth delivery platform. Data from Aim 1 will inform the content and structure of intervention components to be included. During intervention development, two rounds of usability testing will be conducted with 8-10 YMSM, Trans, and gender non-conforming youth to ensure features are usable and the content is understood. Internal beta testing will be performed to assess for full technical functionality.

Specific Aim 3: Evaluate the feasibility, acceptability and preliminary efficacy of PrEP2Prevent with a racially/ethnically diverse sample of 150 (50 Non-Hispanic Whites, 50 Blacks/African American, 50 Latino/Hispanic) YMSM, Trans, gender non-conforming youth, ages 16-26 years. Participants will be randomly assigned in a 1:1 ratio to the intervention app (PrEP2Prevent) or control app (standard of care). Primary outcomes are feasibility, acceptability and preliminary efficacy. Feasibility data will include sources and rates of recruitment/retention, barriers and facilitators to recruitment/retention, engagement with PrEP navigator both in-person and via mHealth platform, as well as paradata on the mHealth platform use (e.g., number of log-ins, time spent, chatroom/text-based discussions). Acceptability will be assessed using a survey with validated measures at intervention completion. Preliminary efficacy will include linkage to PrEP services and PrEP uptake, these data will be collected at baseline and at 3- and 6-months following completion of the intervention. Mediators/moderators will include PrEP self-efficacy, PrEP stigma, and patient activation. The findings from this research will inform further refinements to the intervention and provide estimates of possible intervention effect sizes (group means, SDs) for a future randomized controlled trial (RCT). The funded research is highly significant, timely and innovative. Its innovation lies in the fact that it: a) targets an intervention for YMSM where it is most needed - e.g., on PrEP uptake; b) recognizes that YMSM require tools and support to successfully navigate PrEP services; and c) uses mHealth to deliver the intervention. Moreover, the intervention can be used for both engagement and re-engagement in PrEP uptake for YMSM who cycle in and out of PrEP care. Further, the intervention is potentially easily adaptable and transferable to address other critical PrEP and HIV needs (e.g., uptake of long-acting PrEP and antiretroviral therapy [ART]).

ELIGIBILITY:
Phase 1A:

Inclusion criteria:

* PrEP providers serving YMSM from healthcare and community-based organizations located in Los Angeles County or PrEP Navigators similarly employed by healthcare and community-based organizations that deliver PrEP services to YMSM.
* >18 years of age

Exclusion criteria:

* Not a PrEP provider or navigator serving YMSM from healthcare and community-based organizations located in Los Angeles County
* under 18 years of age

Phase 1B and Phase 2:

Inclusion criteria:

* 16-26 years old
* cisgender male, Trans, gender non-conforming, or identify differently from the gender picked for you at birth
* identify as gay, bisexual, or some other same-sex identity, and/or report having had sex with anyone with a penis during the previous 12 months
* identify as White/Caucasian, Black/African American, Latinx, Asian-Pacific Islander, Indigenous, Native American or mixed-race
* living in the Los Angeles metro area
* have daily access to an iOS/Android smartphone and/or tablet with internet access
* know their HIV status and are HIV negative at time of enrollment.

Exclusion Criteria:

* is younger than or older than 16- to 26-years
* not cisgender male, Trans, gender non-conforming, or identify differently from the gender picked for you at birth
* does not identify as gay, bisexual, or some other same-sex identity, and/or report having had sex with anyone with a penis during the previous 12 months
* does not identify as White/Caucasian, Black/African American, Latinx, Asian-Pacific Islander, Indigenous, Native American or mixed-race
* does not report living in the Los Angeles metro area
* is non-English speaking
* does not have daily access to an iOS/Android smartphone and/or tablet with internet access
* is a person living with HIV
* for Phase 2 only, participants will be excluded if they participated in the Phase 1B focus groups

Phase 3:

Inclusion criteria:

* 16-26 years old
* cisgender male, Trans, gender non-conforming, or identify differently from the gender picked for you at birth
* identify as gay, bisexual, or some other same-sex identity, and/or report having had sex with anyone with a penis during the previous 12 months
* identify as White/Caucasian, Black/African American, Hispanic/Latino/Latinx, or mixed-race
* living in the Los Angeles metro area
* have daily access to an iOS/Android smartphone and/or tablet with internet access
* report having insertive and/or receptive anal sex in the previous 6 months or report a positive STI result in the previous 6 months
* not currently on PrEP and no plan to start/restart PrEP in the following 7 days
* not currently enrolled in another HIV prevention study

Exclusion criteria:

* is younger than or older than 16- to 26-years
* not cisgender male, Trans, gender non-conforming, or identify differently from the gender picked for you at birth
* does not identify as gay, bisexual, or some other same-sex identity, and/or does not report having had sex with anyone with a penis during the previous 12 months
* does not identify as White/Caucasian, Black/African American, Hispanic/Latino/Latinx, or mixed-race
* does not report living in the Los Angeles metro area
* is non-English speaking
* is a person living with HIV (self-reported)
* does not report insertive and/or receptive anal sex in the previous 6 months or does not report a positive STI result in the previous 6 months
* does not have daily access to an iOS/Android smartphone and/or tablet with internet access
* is currently on PrEP or has plans to start/restart PrEP in the following 7 days; and 11) is currently enrolled in another HIV prevention study.

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cismale, Transgender, non-binary
Enrollment: 150 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Formative Research - PrEP Provider and Navigator Interviews | 90 minute one time interview
  16 qualitative interviews with PrEP Providers and Navigators will be recorded and transcribed. Using existing theory or prior research, researchers will begin by identifying key concepts or variables as initial coding categories. MAXQDA will provide support in the coding and the ability to better understand and identify emergent themes and conceptual frameworks through network maps. These maps may include: 1) components most relevant for an intervention; 2) effective strategies for activation, motivation and engagement; 3) attitudes and challenges related to PrEP; 4) differences in needs, challenges and expectations across ethnic groups; and/or 5) most relevant/important mHealth features. The maps will then be analyzed to identify the relationships between constructs related to the PrEP cascade and relevant components of an online PrEP navigation model.
Formative Research - Youth Working Groups | 4 week duration
  Two working groups, each with 6-10 racial/ethnically diverse YMSM, Trans, and gender non-conforming youth will be conducted. Working groups will meet weekly (or bi-weekly) for up to four sessions. Participants will be guided in discussions on a variety of topics, including 1) experiences with perceptions of PrEP; 2) understanding how YMSM, Trans, and gender non-conforming youth access care; 3) factors that impact uptake of and use to PrEP; 4) risk perceptions and health as a priority; 5) preferred modality (mobile app, web-based, online chat/video) and frequency of navigation activities; and 6) strategies to increase patient activation self-efficacy, advocacy, motivations). A baseline survey about personal health, health history and technology will be given to participants before their first session. At the end of each session, a satisfaction survey will be given to participants to fill out.
Pre-Pilot Mobile App Usability Testing | 4 week duration
  Recruitment of 8-10 racial/ethnically diverse YMSM, Trans, and gender non-conforming youth. Study participants will participate in one online focus group session to download and review the app, one virtual session with the live PrEP Navigator in either chat or video conference format, and a one-on-one exit interview with a research staff member about their app feedback. Participants will also be asked to fill out Pre-Test and Post-Test survey measures to assess app feedback and general usability. Members of the working groups will be invited to use PreP2Prevent over a 2-week period acting in the role of participants. Beta testing will allow for a full assessment of both the technical functionality of the mHealth platform, and will help finalize pilot test procedures. This will include engaging with the peer navigator in two "mock" navigation sessions (one text-based and one video-based).
Patient Navigation Feasibility | 6 Months
  Source: Study logs, Post-navigation satisfaction survey Description: # navigation sessions attended/missed, delivery modality (in-person, text, video); # contacts navigator made to schedule each session, # referrals made/attended. Feasibility defined as at least 50% of individuals attending on average >2 sessions over the 3-month intervention period and a mean post-navigation satisfaction survey score of 4 or higher.
Patient Navigation Acceptability | 6 Months
  Source: In-app survey Description: A brief satisfaction assessment (5 questions) will be administered at the end of each navigation session to identify challenges experienced by the participant, the most and least helpful aspects of the session, challenges using the system, satisfaction with information provided, and any additional needs the participant had that the navigator was not able to address.
PrEP Uptake | 6 Months
  Source: Self report Description: PrEP usage quantitative measures at 3 and 6 months
  Source: Ursure Description: Point-of-care rapid urine test of tenofovir as a biological marker of recent (within 48 hours) PrEP use

CONTACTS AND LOCATIONS:
Overall Officials: Michele D Kipke, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers interested in the PrEP2Prevent data can request access to baseline and follow up survey data, specimen collection data and qualitative data from the phase 1 provider interviews in the form of written transcriptions. A publication plan and data use agreement would be reviewed and approved by the PI's prior to sharing any data.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 8/1/2023-7/31/2026
Access Criteria: Describe how to access this data. Email requests can be submitted to the Senior Programs Manager Lindsay Slay at lslay@chla.usc.edu or PI Michele Kipke at mkipke@chla.usc.edu. Templates will be provided for the publication plan and data use agreement.

REFERENCES:
- [Derived] Stocks JB, Calvetti S, Rosso MT, Slay L, Kipke M, Puentes M, Hightow-Weidman LB. Evaluating the Feasibility and Acceptability of a Digital Pre-Exposure Prophylaxis Navigation and Activation Intervention for Racially and Ethnically Diverse Sexual and Gender Minority Youth (PrEPresent): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 29;12:e50866. doi: 10.2196/50866. PMID 37773616

DOCUMENTS (1):
  • Informed Consent Form (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT05281393/ICF_000.pdf